CLINICAL TRIAL: NCT02328430
Title: Comparison of Remote Camera Measures of Lung Function Compared to Standard Spirometry
Brief Title: Feasibility and Validity of Remote Lung Function Assessment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: North Bristol NHS Trust (Other)
Collaborators: University of Bristol (Other)
Responsible Party: Sponsor
Other Study IDs: 3480
Record Dates: First submitted 2014-12-19; First posted 2014-12-31 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Chronic Lung Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Kinnect 3 camera — comparison of Kinnect 3 measures of chest wall movement during standard spirometry

SUMMARY:
Comparison of standard spirometry to non invasive remote lung function measures of chest wall movement using depth camera technology.

DETAILED DESCRIPTION:
This study plans to test a new non invasive way of measuring lung function and compare it to the current method of blowing into a spirometer.

Spirometry is an essential investigation for diagnosis and assessment of severity in people with Chronic Obstructive Pulmonary Disease (COPD) and other respiratory conditions, it is used in every respiratory unit and across primary care. It requires subjects to blow into a tube which measures volume and flow of expired air. It involves specialist equipment and training to perform and interpret. Not all patients are capable of performing spirometry, in particular children, frail, cognitively impaired and those experiencing a flare or exacerbation of symptoms. Remote lung function assessment technology has the potential to enable assessment of lung function in these groups of patients. In the future it is also hoped that it could be used to improve respiratory disease monitoring outside the healthcare environment such as in the patients home.

This new method uses the latest infra-red depth detection cameras to measure chest wall movement. (N.B this does not capture identifiable images). We would like to record participants chest wall movements while blowing into the spirometer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients attending outpatient department in respiratory medicine.
2. Scheduled to undergo spirometry -

Exclusion Criteria:

1. Unable to give informed consent
2. Unable to perform spirometry -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients attending UK secondary care outpatient department in respiratory medicine and how are scheduled to undergo spirometry
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Correlation between change in chest wall depth and Forced Expiratory Volume in 1 second (FEV1) | participants will be followed up for the duration of outpatient visit - on average 3 hours
  Change in lung volume over time (litre per minute)

CONTACTS AND LOCATIONS:
Overall Officials: James W Dodd, MB CHB PhD, Principal Investigator — Academic Clinical Lecturer
Locations (1):
- North Bristol NHS Trust, Bristol, Avon, United Kingdom